CLINICAL TRIAL: NCT02565095
Title: Interaction of Otolith Stimulation and Carotid Baroreflex in Humans
Acronym: OTOBAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 08-128
Record Dates: First submitted 2015-08-10; First posted 2015-10-01 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Carotid Baroreflex measurements (Other)
  Interventions: Procedure: Stimulation of the carotid baroreceptors with a pressure system

INTERVENTIONS:
Procedure: Stimulation of the carotid baroreceptors with a pressure system — In each decubitus, trains of stimuli 8 (-80, -60, -40, -20, 0, 10, 20 and 40 Torr), with a duration of 500 milliseconds each, will be applied using a positive and negative pressure system placed around the neck of the subject.

SUMMARY:
It is well documented that a few days stay in space induces a change in the vestibular-ocular reflex reflecting a reinterpretation of sensory inputs following the disappearance of gravity. If the change of eye reflexes actually the result of a reinterpretation of sensory input, the investigators should also expect to see an alteration of the vestibular-cardiovascular reflexes. The modification of these reflexes may modulate the carotid baroreflex and thus participate in the post-flight cardiovascular deconditioning.

The first objective of this project is to study the carotid baroreflex under different supine (dorsal, ventral and lateral) inducing different otolith stimulation in normal-gravity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, male and / or female aged 18-30 years
* subject affiliated to a social security scheme, agreeing to participate in the study and who provided informed consent.

Exclusion Criteria:

* who participated in a clinical trial within less than the period of exclusion from this project
* with a past or present history of heart disease, vascular, neurological, respiratory, rheumatological, metabolic or otologic.
* pregnant women (dosage beta HCG)
* having taken any medication heart, vascular, neurological, respiratory, rheumatological, metabolic or might interfere on vestibular test results during the two years preceding the experiment.
* smoking or smoking more than 5 cigarettes / day, 1 cigarette / day or 1 pipe / day

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2009-03; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Arterial flow in Common Carotid Artery (EchoDoppler) | baseline
  Measurements of Common Carotid Artery Blood Flow in Cm/s
Arterial flow in Internal Carotid Artery (EchoDoppler) | Baseline
  Measurements of Internal Carotid Artery Blood Flow in Cm/s
Arterial flow in External Carotid Artery (EchoDoppler) | Baseline
  Measurements of External Carotid Artery Blood Flow in Cm/s
Arterial flow in Vertebral Artery (EchoDoppler) | Baseline
  Measurements of Vertebral Artery Blood Flow in Cm/s

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratoire de Physiologie, CHU de Caen, Caen, France